CLINICAL TRIAL: NCT06332937
Title: Complication Following Postmastectomy Breast Reconstruction
Brief Title: Breast Reconstruction
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ung Sik Jin, Professor, Seoul National University Hospital
Other Study IDs: H-2102-079-1197
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Breast Implant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: postmastectomy breast reconstruction — postmastectomy immediate breast reconstruction

SUMMARY:
Complications following postmastectomy breast reconstruction can compromise surgical outcomes and lead to significant morbidity. The aim of this study was to determine factors associated with complication following two-stage implant-based reconstruction

ELIGIBILITY:
Inclusion Criteria:

* Patients who received implant-based breast reconstruction following mastectomy between 2015 and 2020 in Seoul National University Hospital

Exclusion Criteria:

* Patients who received flap surgery simultaneously with implant insertion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Immediate implant-based breast reconstruction following mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection | 7 years
  Number of patients who developed requiring hospitalization-requiring infection

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea